CLINICAL TRIAL: NCT01002404
Title: The Use of Guide Wire in Biliary Cannulation: Angled or Straight Tipped Guide Wire?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hanna Vihervaara, gastrointestinal surgeon, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/180/2009
Record Dates: First submitted 2009-10-05; First posted 2009-10-27 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Deep Biliary Cannulation
Keywords: ERCP; deep biliary cannulation; guide wire cannulation; post-ERCP pancreatitis; Success of deep biliary cannulation; Rate of post-ERCP pancreatitis; Time used to deep biliary cannulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- angled tipped guide wire (Active Comparator): angled tipped guide wire used to deep biliary cannulation
  Interventions: Procedure: angled and straight tipped guide wire
- straight tipped guidewire (Active Comparator): straight guide wire used to deep biliary cannulation
  Interventions: Procedure: angled and straight tipped guide wire

INTERVENTIONS:
Procedure: angled and straight tipped guide wire — Angled or straight tipped guide wire is used in the beginning of deep biliary cannulation in ERCP . If there is no success, other normal procedures (e.g. double wire cannulation and precut) are performed.

SUMMARY:
The purpose of the study is to prospectively evaluate the deep biliary cannulation in ERCP with the angled tipped guide wire or the straight tipped guide wire.

DETAILED DESCRIPTION:
Patients coming to ERCP examination are being divided randomly to two different groups. The deep biliary cannulation is started with predetermined guide wire. If the cannulation does not succeed in two minutes, the procedure is continued as normal.

ELIGIBILITY:
Inclusion Criteria:

* the need for ERCP assessed by a specialist in gastrointestinal surgery

Exclusion Criteria:

* prior sphincterotomy
* age under 18
* age over 90
* contrast media allergy
* inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The success rate of deep biliary cannulation | October 2010

SECONDARY OUTCOMES:
Frequency of post-ERCP pancreatitis | October 2010
time spent to deep biliary cannulation | October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hanna R Vihervaara, Principal Investigator — Turku University Hospital; Juha Grönroos, PhD, Study Director — Turku University Hospital; Paulina Salminen, PhD, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland